CLINICAL TRIAL: NCT00884351
Title: Magnetoencephalography in Absence Seizures
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090125; 09-N-0125
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-06-15

CONDITIONS: Seizures
Keywords: Epilepsy; MEG; Seizures
MeSH Terms: conditions — Seizures; Epilepsy

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* An absence seizure is a type of seizure that usually begins in childhood and goes away by early adulthood. Scientists do not yet know where absence seizures begin in the brain. Some evidence suggests that these seizures begin in the thalamus, a structure deep in the brain, but other studies suggest that they begin in the frontal cortex, at the front part of the brain.
* Magnetoencephalography is a type of brain scanning procedure that is useful in determining information about what happens to the brain during epileptic seizures. Understanding where absence seizures come from may help doctors find new treatments for them.

Objectives:

* To gain a better understanding of which parts of the brain are affected in absence seizures.

Eligibility:

* Patients 7 to 35 years of age who have been diagnosed with absence seizures.

Design:

* Procedures are for research purposes only, not to diagnose or treat a particular medical condition.
* Two outpatient visits to the National Institutes of Health Clinical Center: evaluation and scanning.
* Researchers will evaluate potential participants with a medical history, physical examination, and electroencephalography (EEG). These tests will be performed under another protocol, 01-N-0139.
* Patients will undergo magnetoencephalography (MEG) and magnetic resonance imaging (MRI) of the brain. The study procedures will be performed one time; however, an MEG or MRI scan may need to be repeated for technical reasons. Researchers will not do more than two MEG or MRI scans.
* The MEG will record very small magnetic field changes produced by the activity of the brain. An EEG will be recorded at the same time as the MEG.
* The MRI will use a magnetic field to take pictures of the inside of the brain.
* The MEG will take 3 hours to complete (2 hours for preparation, 1 hour in the scanner). The MRI will take approximately 1 hour.

DETAILED DESCRIPTION:
Objective:

This protocol will test the hypothesis that the 3-Hz spike-wave discharges seen in absence epilepsy originate in the thalamus. We will use an emerging modality, magnetoencephalograpy (MEG), to test this hypothesis.

Study Population:

33 patients with absence seizures.

Design:

This is a non-invasive imaging study that involves a 275-channel whole head MEG recording and a structural MRI for co-registration of MEG data.

Outcome Measure:

The primary outcome measure is the source localization of spike-wave discharges on magnetoencephalography.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age 7-35
  2. Absence of seizures based on clinical and electroenecephalography data. Patients who have other seizure types (myoclonic, generalized tonic-clonic) in addition to absence seizures may be included.
  3. Patients who have other neurologic disorders may be included, as long as they are able to consent/assent.

EXCLUSION CRITERIA:

1. Contraindications to MEG studies (Dental braces, permanent retainers, metal dental caps/crowns/fillings)
2. Contraindications to MRI studies (such as pacemakers, cochlear devices, surgical clips, metallic implants, orthopedic pins, shrapnel, permanent eyeliner, vagus nerve stimulator)
3. Claustrophobia or anxiety disorders exacerbated by MRI
4. Pregnancy
5. Inability to provide consent/assent

Ages: 7 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2009-04-15; Study Completion 2011-06-15

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Avoli M, Gloor P. Role of the thalamus in generalized penicillin epilepsy: observations on decorticated cats. Exp Neurol. 1982 Aug;77(2):386-402. doi: 10.1016/0014-4886(82)90252-7. No abstract available. PMID 7095066
- [Background] Bernasconi A, Bernasconi N, Natsume J, Antel SB, Andermann F, Arnold DL. Magnetic resonance spectroscopy and imaging of the thalamus in idiopathic generalized epilepsy. Brain. 2003 Nov;126(Pt 11):2447-54. doi: 10.1093/brain/awg249. Epub 2003 Aug 5. PMID 12902313
- [Background] Castro-Alamancos MA. Neocortical synchronized oscillations induced by thalamic disinhibition in vivo. J Neurosci. 1999 Sep 15;19(18):RC27. doi: 10.1523/JNEUROSCI.19-18-j0005.1999. PMID 10479720